CLINICAL TRIAL: NCT01605058
Title: Visual Performance Adn Quality of Vision Evaluation After Implantation of a Trifocal Intraocular Lens
Brief Title: Visual Performance With a Trifocal Intraocular Lens
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: BMI Southend Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Agrippa, Optometrist, BMI Southend Hospital
Other Study IDs: TRI 1.1
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the visual performance of a trifocal intraocular lens at distance, near and intermediate viewing, by way of visual acuity measurement, contrast sensitivity.

Patient satisfaction and quality of vision will also be assessed by way of a questionnaire.

DETAILED DESCRIPTION:
Monocular and Binocular Unaided (UCVA) and Best Corrected Visual Acuity (BCVA) will be measured at 6m in LogMAR units under photopic conditions (85cd/m2).

Subjective Refraction will be performed to establish any residual refractive error will for distance, intermediate and near.

Defocus Profiles (visual acuity over imposed defocus) are measured for each patient. The patient observes the 6m LogMAR chart through best distance correction, then defocusing is achieved by the addition of pairs of lenses from +2.00D to -4.00D in 0.50D steps.. The LogMAR acuity will be recorded and the data plotted.

Contrast Sensitivity will be evaluated monocularly under photopic (85cd/m2) conditions and mesopic (4cd/m2) using the Pelli-Robson Contrast Sensitivity Chart.

Near and intermediate performance will be evaluated using the Radner Reading Charts to assess acuity (LogRAD units) and reading speed in photopic conditions 85cd/m2

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70yrs
* Bilateral implantation of a trifocal intraocular lens

Exclusion Criteria:

* existing ocular pathology
* surgical complications
* corneal astigmatism > 1.50DC

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from a private ophthalmology clinic
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M Agrippa, BSc, Principal Investigator — BMI Southend
Locations (1):
- BMI Southend Hospital, Westclifff-on-Sea, Essex, United Kingdom